CLINICAL TRIAL: NCT00786071
Title: A Systematic Metabolic Approach to the Evaluation of Nutrition in Rett Syndrome According to the Cardiorespiratory Phenotype in Dutch Rett Girls
Brief Title: Metabolic Evaluation of Nutrition in Rett Syndrome
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. dr. L.M.G. Curfs, University Hospital Maastricht.
Other Study IDs: MEC 08-2-119; NL25356.068.08 (Other: Medical Ethical Committee University Hospital of Maastricht)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome.; Nutritional status.; Metabolic alterations.
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, serum, dried blood spot, leukocytes, erythrocytes, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rett syndrome girls: The study population consists of a well-defined group of Dutch RTT thirteen girls with complete clinical, molecular and neurophysiological work-up.

SUMMARY:
Rett syndrome (RTT) is an X-linked severe neurodevelopmental disorder. Despite their good appetite, many females with RTT meet the criteria for moderate to severe malnutrition. The pathological mechanism is barely understood. Although feeding difficulties may play a part in this, other constitutional factors as altered metabolic processes are suspected. Irregular breathing is a common clinical feature, reflecting the immaturity of the brainstem in RTT. The primary pathophysiology is a defective control mechanism of carbon dioxide exhalation that leads to chronic respiratory alkalosis or acidosis. We assume that chronic respiratory acidosis or alkalosis causes derangement of the metabolic equilibrium in RTT females with important nutritional consequences.

The aims of this pilot study are to describe the nutritional status of the RTT girls and to examine the consequences of a chronic respiratory acidosis or alkalosis on metabolic processes as a possible cause of impaired nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RTT (meeting consensus diagnostic criteria (Hagberg et al, 2002));
* MECP2-mutation;
* Complete neurophysiological work-up.

Exclusion Criteria:

* Male gender.

Ages: 2 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of a well-defined group of thirteen Dutch RTT girls with complete clinical, molecular and neurophysiological work-up.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
1. What is the nutritional status of the RTT girls? 2. Can metabolic alterations caused by chronic respiratory acidosis or alkalosis be detected? | Once.

CONTACTS AND LOCATIONS:
Overall Officials: Leopold MG Curfs, Professor, Study Director — Maastricht University Medical Center; Eric EJ Smeets, MD, PhD, Study Director — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Reilly S, Cass H. Growth and nutrition in Rett syndrome. Disabil Rehabil. 2001 Feb 15-Mar 10;23(3-4):118-28. doi: 10.1080/09638280150504199. PMID 11247007
- [Background] Oddy WH, Webb KG, Baikie G, Thompson SM, Reilly S, Fyfe SD, Young D, Anderson AM, Leonard H. Feeding experiences and growth status in a Rett syndrome population. J Pediatr Gastroenterol Nutr. 2007 Nov;45(5):582-90. doi: 10.1097/MPG.0b013e318073cbf7. PMID 18030237
- [Background] Rocchigiani M, Sestini S, Micheli V, Pescaglini M, Jacomelli G, Hayek G, Pompucci G. Purine and pyridine nucleotide metabolism in the erythrocytes of patients with Rett syndrome. Neuropediatrics. 1995 Dec;26(6):288-92. doi: 10.1055/s-2007-979776. PMID 8719742
- [Background] Sierra C, Vilaseca MA, Brandi N, Artuch R, Mira A, Nieto M, Pineda M. Oxidative stress in Rett syndrome. Brain Dev. 2001 Dec;23 Suppl 1:S236-9. doi: 10.1016/s0387-7604(01)00369-2. PMID 11738881
- [Background] Viola A, Saywell V, Villard L, Cozzone PJ, Lutz NW. Metabolic fingerprints of altered brain growth, osmoregulation and neurotransmission in a Rett syndrome model. PLoS One. 2007 Jan 17;2(1):e157. doi: 10.1371/journal.pone.0000157. PMID 17237885
- [Background] Julu PO, Engerstrom IW, Hansen S, Apartopoulos F, Engerstrom B, Pini G, Delamont RS, Smeets EE. Cardiorespiratory challenges in Rett's syndrome. Lancet. 2008 Jun 14;371(9629):1981-3. doi: 10.1016/S0140-6736(08)60849-1. No abstract available. PMID 18555901